CLINICAL TRIAL: NCT06360666
Title: Clinical Outcomes in Adult Patients Undergoing Laparoscopic Surgery Under Neuraxial Anesthesia
Acronym: NEURAX
Status: Enrolling by invitation | Type: Observational
Sponsor: Asst Melegnano e Martesana (Other Government)
Responsible Party: Principal Investigator, Davide Vailati, MD, Anesthesiologist, Principal Investigator, Asst Melegnano e Martesana
Other Study IDs: Neurax1
Record Dates: First submitted 2024-03-26; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Mortality; Surgical Complication; Neurological Complication; Respiratory Complication; Cardiovascular Complication; Nephrotoxicity; Metabolic Complication
Keywords: awareness; locoregional anesthesia; general anesthesia; laparoscopic abdominal surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- General Anesthesia: Patients undergoing elective laparoscopic major surgery in general anesthesia
- Loco Regional Anesthesia - Awareness: Patients undergoing elective laparoscopic major surgery using a combined subarachnoid and thoracic epidural anesthesia approach, keeping the patient spontaneously breathing

SUMMARY:
The goal of this observational study is to learn about postoperative mortality and postoperative length of stay outcomes after abdominal laparoscopic major surgery. The main question it aims to answer is:

Does general anesthesia lower complications compared to loco-regional anesthesia (keeping the patient spontaneously breathing and sedated) in laparoscopic abdominal major surgery? Participants are followed for neurological sequelae for 90 days following surgery

DETAILED DESCRIPTION:
BACKGROUND Laparoscopic abdominal surgery has historically required general anesthesia. However, the use of general anesthetics has neurological effects, including the risk of postoperative neurological disorders. Cognitive impairments (amnesia, cognitive delay, postoperative cognitive dysfunction, difficulty in resuming daily activities) occur in variable percentages of patients based on the type and dosage of anesthetics, duration of exposure, cerebral perfusion pressure, baseline cognitive status, and patient age. Mechanical ventilation during general anesthesia often leads to lung atelectasis, compounded by reduced diaphragmatic excursion due to laparoscopic insufflation, potentially impacting tissue oxygenation and leading to postoperative complications. General anesthetics also have negative inotropic and chronotropic effects, affecting tissue perfusion and increasing the risk of neurological and surgical complications and cardiovascular events.

The increasing complexity of surgical techniques and patient comorbidities necessitates exploring alternatives to general anesthesia, particularly for fragile patients undergoing laparoscopic abdominal surgery. Regional anesthesia techniques have been advocated to provide effective anesthesia while minimizing neurological, cardiovascular, and respiratory impacts, thereby improving clinical outcomes and functional recovery.

RATIONALE Given the significant impact of anesthesia on postoperative complications in fragile patients undergoing laparoscopic abdominal surgery, we aim to develop an anesthetic strategy that optimizes clinical and functional outcomes, especially in terms of preserving neurocognitive and respiratory function, by reducing reliance on general anesthetics. This has led us to reconsider regional anesthesia as an alternative during laparoscopic abdominal surgery.

STUDY DESIGN This is a retrospective observational cohort clinical study, monocentric, with analysis of previous months (following acquisition of study consent) and follow-up.

Each patient underwent preoperative evaluation with a standard anesthesiology visit based on national and international guidelines (SIAARTI-ERAS-ESC). Additionally, preoperative neurologic status was assessed using the Mental Test, delirium assessment with NU-Desc, and Frailty Scale. Lung ultrasound assessment was routinely performed on the day of surgery (see attached assessment scores) before the start of anesthesia procedures and again 2 hours after surgery completion. Patients were sedated with non-GABAergic anesthetics, targeting RASS 0/-2.

Data related to procedures performed, anesthetic techniques used, complications, radiological and laboratory reports will be extracted anonymously from the Dedalus O4C, T4Health, and TrackCare applications.

Information, in aggregated form and stratified by type of procedure, will be collected in a Microsoft Excel database and used for subsequent statistical analysis.

FOLLOW-UP At 1 and 3 months, during routine post-operative visits, patients were assessed for neurologic status (Mental Test, delirium assessment with NU-Desc, Frailty Scale). Mortality was assessed at 3 months post-surgery. Patients followed at other centers were contacted by phone to assess neurologic status and mortality.

STATISTICAL ANALYSIS Data were treated anonymously and managed using an electronic Case Report Form (eCRF) developed with the Microsoft Excel platform. Data related to neurologic reassessments during follow-ups are reported in the data collection sheet developed using Microsoft Excel.

Statistical analysis will be performed using MedCalc™ version 20.118 32-bit. Appropriate statistical tests including ANOVA, Chi-square test, and T-test will be used where applicable. Continuous variables will be expressed as mean ± standard deviation, categorical variables as percentages. Variables with a p-value <0.05 will be considered statistically significant.

RESULTS PUBLICATION Publication of study data will occur upon study completion.

ETHICAL/LEGAL ASPECTS

9.1 AC/CE Approval A copy of the patient's informed consent must be submitted to the Ethics Committee (EC) along with the protocol for written approval. Written approval of the protocol and informed consent must be obtained before patient recruitment begins.

EC favorable opinion must be obtained before the trial starts. The researcher should inform the EC of any protocol amendments, which must be approved by the EC.

9.2 Informed Consent All eligible patients will be asked for informed consent to participate in the study.

9.3 Personal Data Handling Personal data collected must comply with the European General Data Protection Regulation (GDPR), Legislative Decree 196/2003 and subsequent amendments, and any other applicable Italian laws for personal data protection ("applicable data protection law").

The Promoter will handle personal data provided in a pseudo-anonymized form in compliance with applicable data protection law.

The Promoter will implement necessary measures to comply with applicable data protection law and implement appropriate technical and organizational measures to ensure GDPR compliance.

The Promoter is responsible for providing Principal Investigators and Research Personnel with necessary information regarding how the Promoter will collect and manage their personal data before such information is provided.

The Promoter ensures correct handling of personal data as required by the GDPR. If a data breach involving personal data is identified, the user must promptly notify other users within 24 hours of becoming aware of the breach. In such cases, the user must cooperate fully to remedy the data breach, fulfill mandatory notification within specified timeframes, and manage any resulting damage.

Data breach involving personal data is defined in articles 33 and 34 of the GDPR.

DATA COLLECTION, MANAGEMENT, AND STORAGE: CRF The study will be conducted in accordance with the Helsinki Declaration and in compliance with good clinical practice norms (Ministerial Decree of Health dated 15/07/1997 and subsequent amendments) and applicable regulatory provisions.

The Promoter will appropriately maintain clinical records and research data in compliance with section 4.9 of ICH-GCP E6, regulatory agency provisions, and institution regulations to ensure patient confidentiality protection. As a participant in a clinical study, the Promoter will allow authorized personnel and regulatory agencies to review (and when permitted by law, copy) clinical records for data quality checks, audits, safety evaluations, and study progress assessments.

Source documents include all information, original records of clinical findings, observations, or other activities necessary for the reconstruction and evaluation of the clinical study. Examples include but are not limited to, medical records, clinical charts, laboratory notebooks, memoranda, patient diaries or assessment lists, drug dispensing records, data recorded by automated instruments, certified copies or transcriptions verified for accuracy and completeness, microfiche, photographic negatives, microfilm or magnetic media, X-ray films, subject cards, and records kept in pharmacies, laboratories, and technical-medical departments involved in the clinical study.

Data collection is the responsibility of personnel at the study center under the supervision of the center's Principal Investigator. The Case Report Form (CRF) is the primary tool for data collection. The researcher should ensure accuracy, completeness, legibility, and timeliness of data entered into the CRF and other relevant data. Data recorded in the CRF, derived from source documents, must match the originals, and any discrepancies should be explained. All required CRF data must be recorded, and any missing data must be explained. Any changes or corrections to a paper CRF must be dated, initialed by the compiler, explained if necessary, and not obscure the original data. The researcher should track changes and corrections made to CRFs.

The researcher/institution should maintain study documents as specified in Essential Documents for Conducting a Clinical Study (ICH-GCP E6, section 8) and as required by regulatory agencies and guidelines. Measures should be taken to prevent accidental or premature destruction of documentation.

Essential documents (written and electronic) should be retained for at least fifteen (15) years from study completion, unless the Promoter provides written authorization to dispose of or retain data for an additional period if permitted by law, regulatory agencies, and/or guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* "ASA physical status">1 (ASA=American Society of Anesthesiologists)
* METs<10 (MET= Metabolic Equivalent)

Exclusion Criteria:

* "ASA physical status"=1
* METs≥10
* patients undergoing laparotomy or emergency surgery, presenting contraindications to central locoregional anesthesia execution (specifically: coagulation disorders, severe spinal malformations, known allergy to local anesthetics, severe aortic stenosis, systemic sepsis, puncture site infection)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients considered for the study will be those undergoing elective laparoscopic major surgery, enrolled in the clinical database for follow-up by the Anesthesia and Intensive Care Unit and General Surgery Unit at the Vizzolo facility - ASST Melegnano e Martesana.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | 90 days
  To determine the rate of postoperative mortality within the two patient cohorts
Morbidity | 90 days
  To determine the number of postoperative length of stay days within the two patient cohorts

SECONDARY OUTCOMES:
Surgical revisions | 90 days
  To correlate the incidence of surgical revisions with the two different anesthesia approaches (general anesthesia and locoregional anesthesia).
organ dysfunctions | 90 days
  To correlate the incidence of organ dysfunctions with the two different anesthesia approaches (general anesthesia and locoregional anesthesia).

CONTACTS AND LOCATIONS:
Locations (1):
- ASST Melegnano e Martesana - Ospedale Vizzolo Predabissi, Vizzolo Predabissi, Milan, Italy

IPD SHARING:
Plan to Share IPD: No